CLINICAL TRIAL: NCT04694716
Title: Determination of Serum Trace Element and Physical Activity Levels in COVID-19 Patients
Brief Title: Determination of Serum Trace Element and Physical Activity Levels in COVID-19
Status: Completed | Type: Observational
Sponsor: Izmir Bakircay University (Other)
Collaborators: Cigli Regional Training Hospital (Other); Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Kadirhan Ozdemir, PT, PhD., Assist. Prof., Izmir Bakircay University
Other Study IDs: 2020-12-141
Record Dates: First submitted 2021-01-03; First posted 2021-01-05 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Covid19
Keywords: Covid-19 (SARS-CoV-2); Serum trace elements; Physical activity
MeSH Terms: conditions — COVID-19; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Covid-19 group (Group I): Patients diagnosed with Covid-19 will be enrolled in this group.
  Interventions: Other: No intervention
- Control group (Group II): Healthy individuals will be enrolled in this group.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention will be applied.

SUMMARY:
The pathogenesis of COVID-19, which is caused by the coronavirus species, which has become a global health problem affecting the lives of billions of people worldwide and is a member of the Betacoronavirus genus, is not fully understood. Although its pathogenesis is thought to be multifactorial, it results in a systemic hyperinflammatory response and associated thromboembolic complications in severe cases. It is thought that some vitamins and nutrients may be beneficial for COVID-19 infected patients due to their anti-inflammatory and antioxidant properties. Vitamins such as A, B, C, D, E and folate; trace elements such as iron, zinc, magnesium, selenium and copper play important roles in supporting both innate and adaptive immune systems, and studies have shown that the trace elements investigated have important roles in COVID-19. For this reason, it is important to investigate the levels of trace elements. In addition, while the disease spreads all over the world, individuals are required to stay at home for a long time against the risk of contamination. Due to these isolation and limitations, physical activity levels decrease in individuals. As reductions in the level of physical activity may cause possible secondary symptoms, another parameter is to determine the physical activity level in order to prevent the potential harmful effects of these protective lifestyle regulations related to COVID-19 and to prevent the restrictions from causing physical inactivity. This study is planning to conduct between January and February 2021 in order to compare the trace element levels in blood samples and physical activity levels of patients with COVID-19 (SARS CoV-2) who applied to Izmir Bakircay University Cigli Training and Research Hospital (Cigli Regional Training Hospital) and hospitalized in the COVID-19 service. It was planned as a prospective, randomized controlled trial. Research data will be obtained from blood samples taken from participants. In addition, data on physical activity levels will be collected through a questionnaire. After analyzing the data obtained from the research with appropriate statistical methods, the data will be evaluated.

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19), also known as Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2), is caused by a coronavirus strain that has become a global health problem by affecting the lives of billions of people worldwide and is a member of the Betacoronavirus genus.

Its clinical presentation can be heterogeneous, ranging from asymptomatic to severe disease, which may be associated with a cytokine storm. The pathogenesis of COVID-19 is not fully understood, but it is likely multifactorial, resulting in a systemic hyperinflammatory response and associated thromboembolic complications in severe cases.

Due to their anti-inflammatory and antioxidant properties, certain vitamins and nutrients may be beneficial for patients infected with COVID-19. Vitamins such as A, B, C, D, E and folate; Trace elements such as iron, zinc, magnesium, selenium and copper have important roles in supporting both innate and adaptive immune systems.

In order to consider an adult to be physically active, it is generally accepted to reach at least 150 minutes of moderate or 75 minutes of high-intensity activity per week, or an equivalent combination of both. Sedentary behavior is defined as wakeful behavior characterized by an energy expenditure of less than 1.5 metabolic equivalent (MET) in positions such as lying, sitting or standing. While the COVID-19 disease spreads all over the world, healthy people are asked to stay at home for a long time against the risk of transmission. As a result, COVID-19 is radically changing the determinants of both behaviors (individual, interpersonal, environmental, regional or national policies and global). Accordingly, it can be said that due to isolation and limitations in regular and joint activities, it can be said that it poses a significant challenge to fulfill physical activity recommendations and reduce sedentary behavior during the stay at home, especially in the first weeks when the chance of finding alternatives to keep the population active even at home is limited. For this reason, individuals are strongly encouraged to engage in physical activity in the home environment by public health advocates to prevent the potential harmful effects of protective lifestyle regulations related to COVID-19 and to prevent the restrictions from causing physical inactivity.

In the light of all this information, in order to contribute to the literature, the aim of this study is to determine the serum trace element levels and physical activity levels of COVID-19 patients immediately before the beginning of COVID-19 treatments and compare with the results of healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of COVID-19 for Group I,
* Not having any chronic diseases for Group II,

Exclusion Criteria:

* Having been taking trace element supplements for the last 2 weeks
* Patients who do not require hospitalization for Group I,
* Patients with a diagnosis of kidney failure and/or heart failure for Group I,
* Patients who are pregnant for Group I

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants in Group I will be included the study from Izmir Bakircay University Cigli Training and Research Hospital (Cigli Regional Training Hospital).
  Participants in Group II will be included the study from community sample.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Levels of serum trace elements parameters | At baseline
  Serum trace elements (zinc, selenium, potassium, sodium, calcium, magnesium, copper) levels will be determined by venous blood samples taken from the participants. Serum trace element levels samples will be analyzed using the atomic absorption spectrophotometry (AAS) method.
Physical Activity Level | At baseline
  International Physical Activity Questionnaire will be used to determine the level of physical activity.

SECONDARY OUTCOMES:
Levels of Routine Blood Samples | At baseline
  Hemogram, levels of vitamin D, Troponin T, D-Dimer, iron, ferritin, C-reactive protein (CRP), lymphocyte/CRP ratio, neutrophil/lymphocyte ratio, levels of procalcitonin, uric acid, chlorine, blood urea nitrogen (BUN) creatine, albumin and bilirubin will be taken from patient files.

CONTACTS AND LOCATIONS:
Locations (1):
- Kadirhan Ozdemir, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No